CLINICAL TRIAL: NCT01742156
Title: Single Blind Randomized Study to Determine the Sensitivity and Specificity of 2 Non-invasive Markers of Early Coronary Disease
Status: Terminated | Type: Observational
Why Stopped: inadequate number of recruita
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nadia Giannetti, Chief of Cardiology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: OPTH-CAD
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: CAD; microangiopathy; patients; more likely; to have tortuosity; of conjunctival vessels
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Presence of coronary disease: All patients with or without coronary disease who are followed in coronary clinics or wards
- coronary disease: Is coronary disease associated with tortuosity of vessels Patients seen in cardiology clinics

SUMMARY:
Diagonal ear lobe crease and microcirculatory disorder in the conjunctiva are both non invasive methods documented in the literature as early signs of coronary artery disease. We wish to study the sensitivity and specificity of both signs by conducting a single blind study involving patients with documented presence or absence of coronary artery disease via angiogram.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 70 years old
* angiogram within past 12 weeks
* stable during post angio period
* willing to provide informed consent

Exclusion Criteria:

* previous eye surgery including cataract surgery
* previous ophthalmologic disorders
* previous surgeries involving ears or ear lobes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients (CCU) and Outpatients (CHF clinic, congenital heart clinic) who have had an angiogram within the past 12 weeks documenting the extent of coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Presence of tortuosity of conjunctival vessels | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Giannetti, MD, Principal Investigator — McGill University
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada